CLINICAL TRIAL: NCT07018947
Title: A Phase II, Randomized, Open-label, National, Multicenter Study Evaluating the Efficacy and Safety of the Combination of Atezolizumab and Bevacizumab as Neoadjuvant Plus Adjuvant Treatment in Hepatocellular Carcinoma (ASPIRE)
Brief Title: Study to Evaluate the Efficacy and Safety of Atezolizumab and Bevacizumab as Neoadjuvant Plus Adjuvant Treatment in HCC
Acronym: ASPIRE
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fundacion Clinic per a la Recerca Biomédica (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-521459-22-00
Record Dates: First submitted 2025-05-27; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Resectable Hepatocellular Carcinoma
Keywords: resectable HCC with high risk of recurrence
MeSH Terms: interventions — atezolizumab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Atezolizumab and Bevacizumab (Experimental): Participants in the atezolizumab plus bevacizumab (Atezo + Bev) arm will receive up to three 3 atezolizumab doses (days 10, 31, 52) and 2 bevacizumab dose (days 10 and 31) until surgery or unacceptable toxicity, whichever occurs first (neoadjuvant therapy).
  The adjuvant therapy with Atezo + Bev will start between 4 and 12 weeks after the resection date, once the participant has fully recovered from the surgery. Participants will receive up to 12 months or 17 cycles of treatment, whichever occurs first, or until disease recurrence or unacceptable toxicity.
  Interventions: Drug: Atezolizumab and Bevacizumab
- Survillance (No Intervention): In Arm Survillance, participants will receive standard of care with no neoadjuvant and adjuvant treatment, undergo surgical resection.

INTERVENTIONS:
Drug: Atezolizumab and Bevacizumab — Participants will receive up to three 3 atezolizumab doses (days 10, 31, 52) and 2 bevacizumab dose (days 10 and 31) until surgery or unacceptable toxicity, whichever occurs first (neoadjuvant therapy).
  The adjuvant therapy with Atezo + Bev will start between 4 and 12 weeks after the resection date, once the participant has fully recovered from the surgery. Participants will receive up to 12 months or 17 cycles of treatment, whichever occurs first, or until disease recurrence or unacceptable toxicity.
  Arms: Atezolizumab and Bevacizumab

SUMMARY:
Study to evaluate the efficacy and safety of the combination of Atezolizumab and Bevacizumab as neoadjuvant plus adjuvant treatment in Hepatocellular Carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form.
2. Age ≥ 18 years at the time of signing Informed Consent Form.
3. Ability to fully comply with the protocol, in the investigator's judgment.
4. Diagnosis of HCC confirmed by histology.
5. HCC that is amenable to R0 surgical resection with curative intent in the opinion of the surgeons and oncologists or hepatologists involved in the care of the participant.
6. HCC at high-risk of recurrence defined by either multifocality, large tumor diameter (>5cm), AFP (alpha-fetoprotein) ≥400ng/mL, poor tumor differentiation, or the presence of microvascular invasion.

   - For patients with tumors between 3-5 cm, a predefined nomogram will be applied, indicating a high prevalence of microvascular invasion with a score >200 points. (Lie et al., 2016).
7. Measurable disease (at least one target lesion) according to RECIST v1.1 as determined by the investigator.
8. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0.
9. Child-Pugh Class A.
10. No evidence of clinically significant portal hypertension (CSPH) or minor CSPH (HVPG <12 mmHg) in candidates for minor resection (fewer than 3 segments). (Galle et al., 2018) Clinically significant portal hypertension (CSPH) can be defined either by its gold standard measurement, a hepatic venous pressure gradient (HVPG) ≥10 mmHg, or by the presence of surrogate markers such as a platelet count <100,000 × 10³/µL combined with splenomegaly.
11. Willing to undergo a tumor biopsy at screening visit.

    - Baseline tumor tissue samples will be collected from all participants by means of a core-needle biopsy performed at study entry. A minimum of two core-needle biopsies are required. If a fresh biopsy is not deemed feasible by the investigator, archival tumor tissue may be submitted, provided the tissue was obtained from a biopsy performed within 3 months prior to enrollment and the patient has not received any anti-cancer therapy, including locoregional liver-directed therapy, since the time of the biopsy. Tumor and normal adjacent tissue specimen will be collected at surgery as fresh snap-frozen and formalin-fixed, paraffin-embedded (FFPE) format. FFPE tissue blocks are preferred, or a minimum of 20 slides must be submitted.
12. No prior locoregional or systemic treatment for HCC.
13. Adequate hematologic and end-organ function, defined by the following laboratory test results:

    * ANC ≥ 1.5 × 109/L (1500/µL) without granulocyte colony-stimulating factor (G-CSF) support.
    * Lymphocyte count ≥ 0.5 × 109/L (500/µL).
    * Platelet count ≥ 75 × 109/L (75,000/µL) without transfusion.
    * Hemoglobin ≥ 90 g/L (9.0 g/dL) without transfusion. Participants must not have required transfusion during screening or within 2 weeks prior to screening to meet this criterion.
    * AST, ALT, and ALP ≤ 5 × upper limit of normal (ULN).
    * Bilirubin ≤ 3 × ULN.
    * Adequate renal function: creatinine clearance by estimated glomerular filtration rate (eGFR) by Modification of Diet in Renal Disease Study (MDRD) formula ≥ 50 mL/min. Participants with creatinine clearance by estimating eGFR by MDRD formula of ≥ 30 mL/min and ≤ 50 mL/min may be enrolled if renal function was stable for ≥ 28 days prior to randomization.
    * Albumin ≥ 28 g/L (2.8 g/dL) without transfusion.
    * For participants not receiving anticoagulation: INR or aPTT ≤ 1.5 × ULN.
14. Documented virology status of hepatitis, as confirmed by screening tests for hepatitis B virus (HBV) and/or hepatitis C virus (HCV):

    * Patients with active HBV must have HBV DNA < 500 IU/mL during screening, must have initiated anti-HBV treatment at least 14 days prior treatment initiation, and must be willing to continue anti-HBV treatment during the study (per local standard of care, e.g., entecavir).
    * Patients with HCV, either with resolved infection (as evidenced by detectable antibody) or chronic infection (as evidenced by detectable HCV RNA), are eligible.
    * For patients with detectable HCV RNA and for whom HCV treatment is considered appropriate by the investigator, treatment should begin no sooner than 6 months following liver resection consistent with AASLD guidelines.
15. Negative HIV test at screening with the following exception:

    - Individuals with a positive HIV test at screening are eligible if they are stable on anti-retroviral therapy, have a CD4 count ≥ 200/mL, and have an undetectable viral load.
16. For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraception.
17. For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraception, and agreement to refrain from donating sperm.

Exclusion Criteria:

1. Presence of extrahepatic disease or macrovascular invasion.
2. Known fibrolamellar HCC, sarcomatoid HCC, mixed cholangiocarcinoma and HCC, or other rare variants of HCC.
3. History of hepatic encephalopathy if clinically significant within one year prior to screening.
4. CSPH in candidates for major resection (more than 3 segments).
5. Moderate or severe ascites.
6. Active co-infection with HBV and HCV (defined as detectable HCV RNA plus positive HBV surface antigen or HBV DNA). Patients with a history of HCV infection but who are negative for HCV RNA by Polymerase Chain Reaction (PCR) will be considered non-infected with HCV.
7. Known active co-infection with HBV and hepatitis D viral infection (HDV).
8. Prior treatment with immune checkpoint blockade therapies, including anti-CTLA-4, anti-PD-1, and anti-PD-L1 therapeutic antibodies.
9. Treatment with investigational therapy within 28 days prior to screening.
10. Untreated or incompletely treated esophageal and/or gastric varices with bleeding or that are at high risk for bleeding. Participants must undergo an esophagogastroduodenoscopy (EGD), and all size of varices (small to large) must be assessed and treated per local standard of care prior to enrollment. Participants who have undergone an EGD within 6 months prior screening do not need to repeat the procedure.
11. A prior bleeding event due to esophageal and/or gastric varices within 6 months prior to screening.
12. Inadequately controlled hypertension, defined as systolic blood pressure (BP) > 150 mmHg and/or diastolic BP > 100 mmHg (average of at least three readings at two or more sessions).

    - Anti-hypertensive therapy to achieve these parameters is allowed.
13. History of hypertensive crisis or hypertensive encephalopathy.
14. Significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to screening.
15. History of hemoptysis (≥ 2.5 mL of bright red blood per episode) within 1 month prior to screening.
16. Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation).
17. Current or recent (≤ 10 days prior to screening) use of aspirin (> 325 mg/day) or treatment with clopidogrel, dipyramidole, ticlopidine, or cilostazol.

    - Chronic use of low dose aspirin (< 325 mg/day) for cardioprotection is allowed.
18. Current or recent (≤ 10 days prior to screening) use of full-dose oral or parenteral anticoagulants or thrombolytic agents for therapeutic (as opposed to prophylactic) purpose.

    * Prophylactic anticoagulation for the patency of venous access devices is allowed provided the activity of the agent results in an INR < 1.5 × ULN and aPTT is within normal limits within 14 days prior to screening.
    * Prophylactic use of low-molecular-weight heparin (LMWH; i.e., enoxaparin 40 mg/day) is allowed. However, the use of direct oral anticoagulant therapies such as dabigatran (Pradaxa®) and rivaroxaban (Xarelto®) are not recommended due to potential bleeding risk. Benefits and risks should be assessed, and caution exercised for use of direct oral anticoagulants.

    The investigator should consider switching to other approved anticoagulants due to the risk of upper GI (gastrointestinal) bleeding in patients with HCC.

    - For prophylactic use of anticoagulants or thrombolytic therapies, the approved dose as described on the local label may be used.
19. History of abdominal or tracheoesophageal fistula, GI perforation, or intra-abdominal abscess within 6 months prior to screening.
20. History of intestinal obstruction and/or clinical signs or symptoms of GI obstruction, including subocclusive or occlusive syndrome related to the underlying disease, or requirement for routine parenteral hydration, parenteral nutrition, or tube feeding prior to screening.
21. Evidence of abdominal free air that is not explained by paracentesis or recent (< 3 months) abdominal surgical procedure.
22. Serious, non-healing, or dehiscing wound, active ulcer, or untreated bone fracture.
23. Grade ≥ 2 proteinuria, as demonstrated by ≥ 2+ protein on dipstick urinalysis and ≥ 1.0 g of protein in a 24-hour urine collection.

    * All patients with ≥ 2+ protein on dipstick urinalysis at screening must undergo a 24-hour urine collection (or an alternative method such as protein/creatinine ratio, per local guidance) for protein and must demonstrate < 1 g of protein in 24 hours.
    * Patients with < 2+ protein on dipstick urinalysis are eligible for the study.
24. History of intra-abdominal inflammatory process within 6 months prior to screening, including but not limited to peptic ulcer disease, diverticulitis, or colitis.
25. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to screening; or abdominal surgery, abdominal interventions or significant abdominal traumatic injury within 60 days prior to screening; or anticipation of need for major surgical procedure, other than potentially curative liver resection, during the study; or non-recovery from side effects of any such procedure.
26. Complete healing from minor surgery (e.g., simple excision, tooth extraction) must have occurred at least 7 days before screening.
27. Chronic daily treatment with a non-steroidal anti-inflammatory drug (NSAID).

    - The occasional use of NSAIDs for the symptomatic relief of medical conditions such as headache or fever is allowed.
28. Serious infection requiring oral or IV antibiotics and/or hospitalization within 4 weeks prior to screening, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia, or any active infection that, in the opinion of the investigator, could impact participant safety.
29. Any serious medical condition or abnormality in clinical laboratory tests that precludes an individual's safe participation in and completion of the study.
30. History of malignancy within 5 years prior to screening, with the exception of the cancer under investigation in this study and malignancies with a negligible risk of metastasis or death (e.g., 5-year OS rate > 90%), such as adequately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, localized prostate cancer, ductal carcinoma in situ, or Stage I uterine cancer.

    * Patients with localized prostate cancer (defined as Stage ≤ pT2c, Gleason score ≤ 7, and prostate-specific antigen (PSA) at prostate cancer diagnosis ≤ 20 ng/mL) treated with curative intent and without PSA recurrence are eligible.
    * Patients with pre-existing low-risk prostate cancer (defined as Stage cT1/T2a, Gleason score ≤ 6, and PSA ≤ 10 ng/mL) who are treatment-naive and undergoing active surveillance are eligible.
    * Patients with malignancies associated with a negligible risk of metastasis or death (e.g., risk of metastasis or death < 5% at 5 years) are eligible provided they meet all of the following criteria:

      * Malignancy treated with expected curative intent (e.g., adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, or ductal carcinoma in situ treated surgically with curative intent)
      * No evidence of recurrence or metastasis by follow-up imaging and any disease-specific tumor markers.
31. Active or history of autoimmune disease or immune deficiency, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, granulomatosis with polyangiitis, Sjögren syndrome, Guillain-Barré syndrome, or multiple sclerosis, with the following exceptions:

    * Patients with a history of autoimmune-related hypothyroidism who are on thyroid-replacement hormone are eligible for the study.
    * Patients with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study.
    * Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met:

      * Rash must cover < 10% of body surface area.
      * Disease is well controlled at baseline and requires only low-potency topical corticosteroids.
      * No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high-potency or oral corticosteroids within the previous 12 months.
32. Pregnancy or breastfeeding, or intention of becoming pregnant during the study.

    - Female participants of childbearing potential must have a negative serum pregnancy test result at screening.
33. Left ventricular ejection fraction (LVEF) < 50% assessed by either transthoracic echocardiogram (TTE) or multiple-gated acquisition (MUGA) scan (TTE preferred test) within 6 months prior to screening.
34. History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins.
35. History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis or evidence of active pneumonitis on screening chest computed tomography (CT) scan.

    - History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
36. Prior allogeneic stem cell or solid organ transplantation.
37. Active tuberculosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2030-11 (Estimated); Study Completion 2030-11 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free survival (RFS) | From randomization to the first documented recurrence of disease or death from any cause, whichever occurs first, assessed up to 5 years.
  Measured by RFS, defined as the time from randomization to the first documented recurrence of disease according to RECIST v1.1 and mRECIST by the investigator's radiology team, or death from any cause (whichever occurs first).

SECONDARY OUTCOMES:
Pathological response | Surgery
  Measured by MPR rate, defined as the proportion of participants with > 70% necrosis of tumor in the tumor bed at the time of surgery, as assessed by central pathological review.
Pathological response | Surgery
  Measured by complete pathological response (pCR) rate, defined as the proportion of participants with an absence of residual tumor at the time of surgery, as assessed by central pathological review.
Overall Survival (OS) | From randomization to death from any cause, assessed up to 5 years.
  Measured by OS, defined as the time from randomization to death from any cause.
Efficacy of neoadjuvant with atezolizumab plus bevacizumab treatment combinations | From randomization to predefined event or death, whichever came first, assessed up to 5 years.
  Measured by Event-free survival (EFS), defined as time from randomization to predefined event, that may include disease progression/toxicity precluding surgery, relapse [ both assessed according to RECIST v1.1 and mRECIST by the investigator's radiology team] or death.
Efficacy of neoadjuvant with atezolizumab plus bevacizumab treatment combinations | Pre-Surgery visit
  Measured by objective response rate (ORR), defined as the proportion of participants with a radiological CR or PR prior to surgery, as determined by the investigator according to RECIST v1.1 and HCC mRECIST. Responses will be assessed and determined according to RECIST v1.1 and HCC mRECIST but are not required to be confirmed by subsequent imaging assessments.
Efficacy of neoadjuvant with atezolizumab plus bevacizumab treatment combinations | Surgery
  Measured by R0 resection rate (proportion of resected participants obtaining an R0 resection). R0 resection is defined as a microscopically margin-negative resection, in which no tumor (gross or microscopic) remains in the primary tumor bed.
Safety and tolerability of neoadjuvant + adjuvant atezolizumab and bevacizumab treatment combinations. | From randomization to last follow-up visit, an averago of 2-5 years.
  Measured by the incidence, nature, and severity of adverse events, serious adverse events, and immune-related adverse events (severity determined according to NCI CTCAE v5.0).
Surgical feasibility in participants receiving neoadjuvant immunotherapy-based treatment combinations | Surgery
  Measured by proportion of participants with delayed or canceled surgery (defined as > 28 days from surgical restaging visit), as well as length of surgical delay, duration of surgery, surgical approach and extent of surgery.
Surgical outcomes in participants receiving neoadjuvant immunotherapy-based treatment combinations | Surgery
  Measured by proportion of participants with length of hospital stays, intraoperative blood loss, and need for intraoperative blood transfusion.
Surgical morbidity in participants receiving neoadjuvant immunotherapy-based treatment combinations | Surgery
  Measured by proportion of participants with length of hospital stays, intraoperative blood loss, and need for intraoperative blood transfusion.
Surgical mortality in participants receiving neoadjuvant immunotherapy-based treatment combinations | Surgery
  Measured by proportion of participants with length of hospital stays, intraoperative blood loss, and need for intraoperative blood transfusion.
Outcomes, morbidity, and mortality in participants receiving neoadjuvant immunotherapy-based treatment combinations. | Post-Surgery visit and from visit 8 to the last visit
  Measured by post-operative surgical complication rates according to the Clavien-Dindo surgical classification. Clinically relevant complications are defined as Clavien-Dindo Grade ≥ IIIa.
Mortality in participants receiving neoadjuvant immunotherapy-based treatment combinations | 90 days after the surgery visit
  Measured by post-operative mortality, defined as death within 90 days after surgery.

CONTACTS AND LOCATIONS:
Locations (13):
- Spain (13):
  - Complejo Hospitalario Universitario de Santiago de Compostela, Santiago de Compostela, A Coruña
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitari de Bellvitge, Barcelona, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital Universitario Reina Sofía, Córdoba, Cordoba
  - Hospital Universitari Josep Trueta, Girona, Girona
  - Hospital General Universitario Gregorio Marañón, Madrid, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid, Madrid
  - Hospital Universitario Virgen de la Victoria, Puerto de la Torre, Málaga
  - Hospital Universitario y Politécnico La Fe, Valencia, Valencia
  - Hospital Universitario de Cruces, Barakaldo, Vizcaya